CLINICAL TRIAL: NCT02046382
Title: Randomized Control Trial of IV Acetaminophen for Post Cesarean Delivery Pain Relief
Brief Title: RCT (Randomized Controlled Trial) of IV Acetaminophen for Post Cesarean Pain Relief
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 13068
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-02

CONDITIONS: Cesarean Section; Pain, Postoperative
Keywords: IV Acetaminophen; Cesarean Section; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Acetaminophen (Experimental): Subjects will receive a 1000mg dose of IV acetaminophen in 100mL solution every 8 hours for 48 hours. The first dose will be administered intraoperatively following delivery of the baby. A total of 6 doses will be given.
  Interventions: Drug: IV Acetaminophen
- Normal Saline (Placebo Comparator): Subjects will receive a 100mL dose of saline every 8 hours for 48 hours. The first dose will be administered intraoperatively following delivery of the baby. A total of 6 doses will be given.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IV Acetaminophen — 1000mg dose of IV acetaminophen in 100mL solution every 8 hours for 48 hours. The first dose will be administered intraoperatively following delivery of the baby. A total of 6 doses will be given.
  Other Names: Ofirmev
  Arms: IV Acetaminophen
Drug: Placebo — 100 mL of Normal Saline every 8 hours for 48 hours. The first does will be administered intraoperatively following delivery of the baby. A total of 6 doses will be given.
  Other Names: Normal Saline
  Arms: Normal Saline

SUMMARY:
This study is being done to evaluate the scheduled use of intravenous (IV) acetaminophen among cesarean section patients. The study hopes to find out if patients who receive scheduled IV acetaminophen for 48 hours following delivery have lower self-reported pain scores and use less narcotic pain medication than patients who do not receive IV acetaminophen.

DETAILED DESCRIPTION:
See Brief Summary

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Scheduled cesarean section delivery
* Patient of TriHealth's Faculty Medical Center or Tri-State Maternal Fetal Medicine Associates
* Singleton pregnancy
* Term delivery (greater than or equal to 37 weeks)
* Spinal/epidural anesthesia with epidural analgesia (duramorph)
* Use of pfannenstiel incision

Exclusion Criteria:

* Weight less than 50 kg
* Allergy to study drugs (acetaminophen, oxycodone, duramorph, NSAIDS)
* Multiple gestation pregnancy
* Cesarean section for pre-term delivery (less than 37 weeks)
* Fetal anomalies
* Inability to use epidural duramorph at time of procedure
* General anesthesia used
* Vertical skin incision
* Opioid addiction
* Liver dysfunction (hepatitis, HELLP (hemolysis, elevated liver enzymes, and low platelet count), preeclampsia)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Lambers, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- TriHealth Good Samaritan Hospital, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Altenau B, Crisp CC, Devaiah CG, Lambers DS. Randomized controlled trial of intravenous acetaminophen for postcesarean delivery pain control. Am J Obstet Gynecol. 2017 Sep;217(3):362.e1-362.e6. doi: 10.1016/j.ajog.2017.04.030. Epub 2017 Apr 25. PMID 28455085

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV Acetaminophen | Normal Saline
Started | 65 | 67
Completed | 57 | 47
Not Completed | 8 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Acetaminophen | Normal Saline | Total
Number analyzed (Participants) | 57 | 47 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (6.0) | 29.6 (6.1) | 29.6 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 47 | 104
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 33 | 27 | 60
  Race: African American | 21 | 19 | 40
  Race: Multiracial | 2 | 1 | 3
  Race: Other | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57 | 47 | 104

OUTCOME MEASURES:

1. Primary Outcome: Total Oxycodone (mg)
Description: Total oxycodone (mg) for breakthrough pain during inpatient stay
Time Frame: approximately 2 - 7 days
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | IV Acetaminophen | Normal Saline
Number analyzed (Participants) | 57 | 47
mg | 47.0 (39.1) | 65.0 (46.2)

2. Secondary Outcome: Number of Participants With Narcotic Associated Side Effects
Description: Only outcome for nausea/emesis is reported.
Time Frame: 2-7 days
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen | Normal Saline
Number analyzed (Participants) | 57 | 47
Participants | 17 | 9

3. Secondary Outcome: Length of Stay
Description: Length of hospital stay (admission to discharge) will be collected.
Time Frame: 2-7 days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | IV Acetaminophen | Normal Saline
Number analyzed (Participants) | 57 | 47
hours | 78 [74 to 95] | 78 [75 to 98]

4. Other Pre Specified Outcome: Total Amount of Ibuprofen During Inpatient Stay
Description: Patients will have access to ibuprofen for mild to moderate pain. The amount consumed during inpatient stay will be collected.
Time Frame: 2-7 days
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | IV Acetaminophen | Normal Saline
Number analyzed (Participants) | 57 | 47
mg | 4786 (2333) | 5260 (1915)

ADVERSE EVENTS:
Arm/Group | IV Acetaminophen | Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/67
Other Adverse Events (participants affected / at risk) | 0/65 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes